CLINICAL TRIAL: NCT02663557
Title: Evaluating the Influence of Day-to-day Blood Pressure Variation in Acute Ischemic Stroke on Adverse Outcomes in Long-term Post-stroke Followup
Brief Title: The Influence of day-to Day BPV on Long-term Adverse Outcomes in Patients Ischemic Stroke
Status: Completed | Type: Observational
Sponsor: Zhu Shi (Other Government)
Responsible Party: Sponsor-Investigator, Zhu Shi, deputy director of neurology department, Dongguan People's Hospital
Organization: Dongguan People's Hospital (Other Government)
Other Study IDs: 2008105150027; 2008105150027 (Other: dongguan sci and tech bureau); A2013836 (Other Grant/Funding Number: guangdong province medical science and research fund)
Record Dates: First submitted 2016-01-21; First posted 2016-01-26 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Stroke
Keywords: stroke, blood pressure, prognosis
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- non-hypertension with lower BPV: patients meeting to flowing two criteria: 1. mean SBP<140 mmHg; 2. Systolic blood pressure-coefficient variation (SBP-CV) < Median SBP-CV
- non-hypertension with higher BPV: patients meeting to flowing two criteria: 1. mean SBP< 140 mmHg; 2. SBP-CV > Median SBP-CV
- hypertension with lower BPV: patients meeting to flowing two criteria: 1. mean SBP> 140 mmHg; 2. SBP-CV < Median SBP-CV
- hypertension with higher BPV: patients meeting to flowing two criteria: 1. mean SBP> 140 mmHg; 2. SBP-CV > Median SBP-CV

SUMMARY:
Stroke is one of the most devastating disorder worldwide. Hypertension has been confirmed to be a major modifiable risk factor for stroke.Even the casual visit hypertension has been managed ideally,there is still surplus risk for stroke re-attack.The purpose of this study is to explore whether variation of 24-hour ambulatory and visit-to-visit blood pressure variability (BPV) contribute to recurrent stroke.

DETAILED DESCRIPTION:
System hypertension has been reported to play the most important role in the development of stroke,and the anti-hypertension therapy is regarded as the cornerstone for stroke secondary prevention. However, even though some proper measures have been taken,there is still surplus risk for recurrent stroke. Recently the variation of system blood pressure has been focused as the candidate of another risk factor.Up to date,this hypothesis remains an intense debate and few studies has been done to clarify it.Besides, the definition of BPV and measurement of BPV parameters are still beyond conformity.In the current study, the long-term and short-term BPV will be taken respectively for patients with prior stroke. Bsed on these parameters, the cohort will be followed up for average 2 years. The predefined outcome include composite cardiovascular events, neuropsychiatric wording, and mortality during followup.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* comorbidity of dementia ( including AD, PDD, FTLD, VaD and so on )
* coexisting severe systematic diseases on admission such as acute coronary syndrome, malignant tumor, plasma dialysis therapy for renal failure, cirrhosis, rheumatic disease that would influence mortality.
* discharge with severe sequelae with mRS>5

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with acute ischemic stroke, which should be verified by define radiological evidences and acute onset of clinical manifestations.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
mortality | 12 months
  all cause death

SECONDARY OUTCOMES:
macrovascular events | 12 months
  stroke, including recurrent ischemic stroke and intra-cerebral hemorrhage, coronary artery events and peripheral artery occlusion
microvascular events | 12 months
  cognition and psychological decline

OTHER OUTCOMES:
non-cardiovascular events | 12 months
  fall,frature and other unexpected adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Zhu Shi, MD,PhD, Study Chair — dongguan peoples' hospital
Locations (1):
- Dongguan Peoples' Hospital, Dongguan, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
The data will not be shared with respect to the privacy of patients info.